CLINICAL TRIAL: NCT03927222
Title: I-ATTAC: Improved Anti-Tumor Immunotherapy Targeted Against Cytomegalovirus in Patients With Newly-Diagnosed WHO Grade IV Unmethylated Glioma
Brief Title: Immunotherapy Targeted Against Cytomegalovirus in Patients With Newly-Diagnosed WHO Grade IV Unmethylated Glioma
Acronym: I-ATTAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Resource shortage
Sponsor: Mustafa Khasraw, MBChB, MD, FRCP, FRACP (Other)
Responsible Party: Sponsor-Investigator, Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00090683
Record Dates: First submitted 2019-04-19; First posted 2019-04-25 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Dendritic cells; Temozolomide; Tetanus; Khasraw; Immunotherapy; Vaccine
MeSH Terms: conditions — Glioblastoma; Tetanus | interventions — Temozolomide; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Intervention Model Description: Newly-diagnosed WHO Grade IV glioma patients with their tumor resected and found to be MGMT unmethylated will be accrued to this study before the standard of care chemoradiation with the goal of treating with dose-intensified TMZ and pp65 loaded dendritic cell vaccine after completion of the standard of care chemoradiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DC vaccination with Td preconditioning and GM CSF (Experimental): This single-arm phase II study will assess the impact of tetanus pre-conditioning and adjuvant GM-CSF on overall survival of newly diagnosed glioblastoma (GBM) patients who have undergone definitive resection, are unmethylated, and completed standard temozolomide and radiation treatment. All enrolled patients will undergo a leukapheresis for the generation of DCs. Patients will then receive approximately 6 weeks of standard of care radiation therapy (RT) and concurrent TMZ. A single post-RT cycle of dose intensified TMZ (100 mg/m2/day for 21 days) will then be given. On day 23 (± 2 days) of the cycle, patients will receive the first of 3 pp65 DC vaccines every 2 weeks. All patients will receive up to a total of 10 DC vaccines
  Interventions: Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs containing GM CSF; Drug: Temozolomide; Biological: Tetanus-Diphtheria Toxoid (Td); Biological: GM-CSF; Biological: 111-Indium-labeling of Cells for in vivo Trafficking Studies

INTERVENTIONS:
Biological: Human CMV pp65-LAMP mRNA-pulsed autologous DCs containing GM CSF — 2x10^7 human CMV pp65-LAMP mRNA-pulsed autologous DCs are given intradermally and bilaterally at the groin site (divided equally to both inguinal regions). Patients will receive up to a total of 10 DC vaccines.
  Other Names: CMV-specific dendritic cell vaccine; DCs
Drug: Temozolomide — Temozolomide is a chemotherapy drug given to all enrolled patients at the post-RT clinic visit as dose-intensified TMZ (100 mg/m2/day for 21 days).
  Other Names: Temodar; TMZ; Temodal
Biological: Tetanus-Diphtheria Toxoid (Td) — Before the first DC vaccination, patients will receive 0.5 mL of Td (tetanus and diphtheria toxoids adsorbed) intramuscularly into the deltoid muscle to ensure adequate immunity to the tetanus antigen. Prior to pp65 DC vaccination #4,(3±1) weeks after leukapheresis 2 the vaccine site will receive a pre-conditioning intradermal injection of Td (1 flocculation unit (Lf), in 0.3 mL of saline for a total of 0.4 mL).
  Other Names: Td pre-conditioning; Td toxoid
Biological: GM-CSF — Granulocyte macrophage-colony stimulating factor (GM-CSF) is a sterile, white, preservative-free lyophilized powder in a vial containing 250 mcg that will be reconstituted in 0.5 mL of sterile water for injection and used as an adjuvant with the DC vaccine.
  Other Names: LEUKINE®; Sargramostim
Biological: 111-Indium-labeling of Cells for in vivo Trafficking Studies — 111-In-labeled DCs are 2 x 10^7 pp65-LAMP mRNA loaded mature DCs labeled with 111-In (50 μCi / 5 x 10^7 DCs) and given i.d. as the fourth vaccine. In up to 16 patients, the fourth vaccine will be labeled with 111-In (50 μCi / 5 x 10^7 DCs) prior to injection.

SUMMARY:
This single-arm phase II study will assess the impact of tetanus pre-conditioning and adjuvant Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) on overall survival of patients newly diagnosed with World Health Organization (WHO) Grade IV glioblastoma who have undergone definitive tumor resection, are cytomegalovirus (CMV) positive and unmethylated, and completed standard temozolomide (TMZ) and radiation treatment. After completion of the standard of care radiotherapy with concurrent TMZ, patients will receive 1 cycle of dose-intensified TMZ followed by pp65-loaded dendritic cell (DC) vaccination beginning on day 23.

DETAILED DESCRIPTION:
Approximately 64 patients with resected, newly-diagnosed WHO Grade IV glioma who are CMV positive and in which the Methylguanine Methyltransferase (MGMT) is not methylated will be accrued to this study before standard of care radiation therapy (RT) and concurrent TMZ, with the goal of treating 48 patients with dose-intensified temozolomide and pp65 loaded dendritic cell vaccine after completion of standard RT and TMZ.

All enrolled patients will undergo a leukapheresis for the generation of DCs. Patients will then receive approximately 6 weeks of the standard of care radiation therapy (RT) and concurrent TMZ at a standard targeted dose of 75 mg/m2/day. For patients whose initial leukapheresis yields less than 3 vaccines, repeat leukapheresis may be obtained. At the post-RT clinic visit, a single post-RT cycle of dose-intensified TMZ (100 mg/m2/day for 21 days) will be given. On day 23 (± 2 days) of the cycle, patients will receive the first of 3 pp65 DC vaccines. Vaccines #1-3 will be given every two weeks (± 2 days). All patients will receive up to a total of 10 DC vaccines, with vaccines administered every 35 days (± 7 days) after the third vaccine, given bilaterally at the groin site unless progression occurs with no further cycles of TMZ. DC vaccines will be given intradermally (i.d.) and divided equally to both inguinal regions. Before the first DC vaccination, patients will receive 0.5 mL of Td (tetanus and diphtheria toxoids adsorbed) intramuscularly into the deltoid muscle to ensure adequate immunity to the tetanus antigen. Patients will undergo leukapheresis again for immunologic monitoring with a specific assessment of baseline antigen-specific cellular and humoral immune responses if needed for further DC generations 14 (± 2) days after vaccine #3. Prior to pp65 DC vaccination #4,(3±1) weeks after leukapheresis 2, the vaccine site will receive a pre-conditioning intradermal injection of Td. Up to 16 patients will receive 111-Indium labeled DCs at the 4th vaccine followed by SPECT/CT imaging immediately, and at 1 and 2 days after injections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Newly diagnosed World Health Organization (WHO) Grade IV Glioma with definitive resection prior to the consent, with a residual radiographic contrast enhancing disease on the postoperative computed tomography (CT) or Magnetic Resonance Imaging (MRI) of <1 cm in maximal diameter in any plane.
* Able to receive standard of care radiation and chemotherapy for approximately 6 weeks duration and of more than 54 Gray (GY)
* MRI post radiation therapy (RT) does not show progressive disease outside the radiation field
* Enough tumor tissue available for determination of methylguanine-DNA methyltransferase (MGMT) gene promoter status (must be unmethylated) or prior pathology report available confirming MGMT gene promoter status
* Cytomegalovirus (CMV) Seropositive
* Karnofsky Performance Status (KPS) of ≥ 70%
* Hemoglobin ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥ 1,000 cells/µl, platelets ≥ 100,000 cells/µl prior to starting TMZ cycle 1 (patient must meet these criteria within 4 weeks after the end of XRT/TMZ to be eligible)
* Serum creatinine ≤ 3 times institutional upper limit of normal (ULN) for age, aspartate aminotransferase (AST) ≤ 3 times institutional upper limit of normal for age
* Bilirubin ≤ 1.5 times upper limit of normal prior to starting TMZ cycle 1 (Exception: Patient has known Gilbert's Syndrome or patient has suspected Gilbert's Syndrome, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
* Signed informed consent approved by the Institutional Review Board
* Female patients must not be pregnant or breastfeeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intrauterine device [IUD; only hormonal], sexual abstinence or vasectomized partner) during the trial and for a period of > 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have a negative serum pregnancy test within 48 hours prior to first study procedure (leukapheresis).
* Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, intrauterine devices (IUDs) [only hormonal], sexual abstinence or prior vasectomy) during the trial and for a period of > 6 months following the last administration of trial drugs.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
* Patients with known potentially anaphylactic allergic reactions to gadolinium- diethylenetriamine penta-acetic acid (DTPA).
* Patients who cannot undergo MRI or SPECT due to obesity or to having certain metal in their bodies (specifically pacemakers, infusion pumps, metal aneurysm clips, metal prostheses, joints, rods, or plates).
* Patients with evidence of tumor in the brainstem, cerebellum, or spinal cord, radiological evidence of multifocal disease, or leptomeningeal disease.
* Severe, active comorbidity, including any of the following:

  1. Unstable angina and/or congestive heart failure requiring hospitalization;
  2. Transmural myocardial infarction within the last 6 months;
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study initiation;
  4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness r requiring hospitalization or precluding study therapy;
  5. Known hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
  6. Known Human Immunodeficiency Virus (HIV) and Hepatitis C positive status;
  7. Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy;
  8. Active connective tissue disorders, such as lupus or scleroderma that, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity.
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin. (Treatment with tamoxifen or aromatase inhibitors or other hormonal therapy that may be indicated in the prevention of prior cancer disease recurrence, are not considered current active treatment.)
* Patients are not permitted to have had any other conventional therapeutic intervention other than steroids prior to enrollment outside of the standard of care chemotherapy and radiation therapy. Patients who receive previous inguinal lymph node dissection, radiosurgery, brachytherapy, or radiolabeled monoclonal antibodies will be excluded
* Current, recent (within 4 weeks of the administration of this study agent), or planned participation in an experimental drug study.
* Known history of autoimmune disease (with the exceptions of medically-controlled hypothyroidism and Type I Diabetes Mellitus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/
- See also: Duke Health — https://www.dukehealth.org/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
Started | 6
Completed | 0
Not Completed | 6
Not completed — Progression | 3
Not completed — CMV testing results inconclusive | 1
Not completed — Unable to generate enough vaccines | 1
Not completed — Early study termination | 1

BASELINE CHARACTERISTICS:
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS) of Subjects Receiving Td Pre-conditioning With GM-CSF
Description: Time in months from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up has OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: duration of the study (up to 3 years and 4.5 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
Number analyzed (Participants) | 6
months | 17.4 [13.3 to NA] — No not enough failure times to estimate the upper bound.

2. Secondary Outcome: Migration and Survival From Vaccine 4
Description: The Cox proportional hazards model will assess the impact of migration on survival after vaccine #4. Migration is defined as the maximum percentage of 111In-labeled dendritic cells (DCs) reaching inguinal nodes during the 48 hours after the 4th vaccination. The hazard ratio associated with a 1-unit change in migration will be estimated with 95% confidence intervals.CSF to site-draining inguinal lymph nodes after Td pre-conditioning and survival after vaccine # 4.
Time Frame: 5 years
Population: Data not collected.
Groups:
- DC Vaccination With Td Preconditioning and GM CSF: Human CMV pp65-LAMP mRNA-pulsed autologous DCs (dendritic cells) containing GM CSF: 2x10^7 human CMV pp65-LAMP mRNA-pulsed autologous DCs are given intradermally and bilaterally at the groin site (divided equally to both inguinal regions). Patients will receive up to a total of 10 DC vaccines.
  Temozolomide: Temozolomide is a chemotherapy drug given to all enrolled patients at the post-RT clinic visit as dose-intensified TMZ (100 mg/m2/day for 21 days).
  Tetanus-Diphtheria Toxoid (Td): Before the first DC vaccination, patients will receive 0.5 mL of Td (tetanus and diphtheria toxoids adsorbed) intramuscularly into the deltoid muscle to ensure adequate immunity to the tetanus antigen. Prior to pp65 DC vaccination #4,(3±1) weeks after leukapheresis 2 the vaccine site will receive a pre-conditioning intradermal injection of Td (1 flocculation unit (Lf), in 0.3 mL of saline for a total of 0.4 mL).
  GM-CSF: Granulocyte macrophage-colony stimulating factor (GM-CSF) is a sterile, white, preservative-free lyophilized powder in a vial containing 250 mcg that will be reconstituted in 0.5 mL of sterile water for injection and used as an adjuvant with the DC vaccine.
  111-Indium-labeling of Cells for in vivo Trafficking Studies: 111-In-labeled DCs are 2 x 10^7 pp65-LAMP mRNA loaded mature DCs labeled with 111-In (50 μCi / 5 x 10^7 DCs) and given i.d. as the fourth vaccine. In up to 16 patients, the fourth vaccine will be labeled with 111-In (50 μCi / 5 x 10^7 DCs) prior to injection.
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
Number analyzed (Participants) | 0

3. Secondary Outcome: Chemokine (C-C Motif) Ligand 3 (CCL3) and Survival From Vaccine 4
Description: The Cox proportional hazards model will assess the impact of CCL3 on survival post-vaccine 4. The hazard ratio associate with a 1-unit increase in CCL3 will be estimated with 95% confidence intervals
Time Frame: 5 years
Population: Data not collected.
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
Number analyzed (Participants) | 0

4. Secondary Outcome: Polyfunctionality and Survival From Vaccine 4
Description: Cox proportional hazards model will assess the association between fold change increase between baseline and the leukapheresis 2 in the frequency of pp65 antigen-specific CD8+ T cells producing three or more cytokines (IFNγ, CCL3, IL-2, TNFα, CD107a), and survival post-vaccine 4. The hazard ratio associate with a 1-unit fold change in polyfunctionality will be estimated with 95% confidence intervals.
Time Frame: 5 years
Population: Data not collected.
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
Number analyzed (Participants) | 0

5. Secondary Outcome: Maximum Peak Increase From Vaccine 1 in Percent Regulatory T Cells (TReg) of CD4+ T Cells
Description: The mean difference in TRegs between vaccine 1 and the maximum measured level post-vaccine 1 will be reported.
Time Frame: 1 year
Population: Data not collected.
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Unacceptable Toxicity
Description: An unacceptable toxicity is defined as any grade 3 or greater toxicity that is possibly, probably, or definitely attributed to the pre-conditioning agent Td or pp65 DC vaccine that does not resolve to baseline within 3 weeks; any Grade 3 hypersensitivity reactions or autoimmune toxicity requiring steroids or hormone replacement; , and is not due to progressive disease, or any life-threatening event not attributable to concomitant medication, co-morbid event, or disease progression. Toxicities will be graded according to the National Cancer Institute Common Toxicity Criteria of Adverse Events (NCI CTCAE) version 5 criteria.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Duration of the study (up to 3 years and 4.5 months)
Arm/Group | DC Vaccination With Td Preconditioning and GM CSF
All-Cause Mortality (participants affected / at risk) | 5/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DC Vaccination With Td Preconditioning and GM CSF (N=6)
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 2
Blurred vision (Eye disorders) | 1
Cholesterol high (Investigations) | 1
Constipation (Gastrointestinal disorders) | 2
Creatinine increased (Investigations) | 1
Depression (Psychiatric disorders) | 2
Dizziness (Nervous system disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 2
Ear pain (Ear and labyrinth disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 2
Fatigue (General disorders) | 5
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
General disorders and administration site conditions - Other, specify (General disorders) | 1
Headache (Nervous system disorders) | 4
Hearing impaired (Ear and labyrinth disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Injection site reaction (General disorders) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Insomnia (Psychiatric disorders) | 1
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Memory impairment (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Urinary tract infection (Infections and infestations) | 2
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT03927222/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT03927222/ICF_000.pdf